CLINICAL TRIAL: NCT01985412
Title: Genome Transplant Dynamics: Non-Invasive Sequencing-Based Diagnosis of Rejection
Acronym: GTD
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Kaiser Foundation Research Institute (Other)
Responsible Party: Principal Investigator, Kiran Khush, Kiran Khush, MD, MAS, FACC, Stanford University
Other Study IDs: 17666
Record Dates: First submitted 2013-05-28; First posted 2013-11-15 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Cardiac Transplant Rejection; Lung Transplant Rejection
Keywords: Rejection; Transplant; Cardiac; Pulmonary; Heart; Lung; Cell-Free DNA; cfDNA; Cell; Free; DNA; Biopsy; Non-Invasive
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A single whole blood specimen from both the donor and recipient of the organ prior to transplant. Additionally, blood samples are taken post-transplant at specified timepoints and spun down into a plasma, buffycoat layer. The plasma and buffycoat are retained while the rest is discarded.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Adult Heart Transplant Recipients: Patients >18 yrs old that received a heart-only transplant and are followed at Stanford Hospital
- Pediatric Heart Transplant Recipients: Patients <18 yrs old that received a heart-only transplant and are followed at Lucile Packard Hospital
- Adult Lung Transplant Recipients: Patients >18 yrs old that received a lung-only transplant and are followed at Stanford Hospital
- Pediatric Lung Transplant Recipients: Patients <18 yrs old that received a lung-only transplant and are followed at Lucile Packard Hospital
- Kaiser Adult Heart Transplant Recipients: Patients >18 yrs old that received a heart-only transplant at Stanford Hospital but are followed at Kaiser Permanente in Santa Clara

SUMMARY:
The purpose of this study is to determine whether shotgun sequencing technology, which can be used to detect donor DNA in recipient plasma, can be used as a rapid, accurate, non-invasive method to detect Acute Cellular Rejection (ACR) after heart transplantation. Currently, all heart transplant recipients undergo invasive heart biopsies to diagnose ACR. Thus, there is an ongoing need to monitor patients for the development of acute and chronic rejection, with the primary goal of non-invasive early detection and treatment to prevent organ damage.

DETAILED DESCRIPTION:
Previous attempts to develop a non-invasive marker of graft rejection have focused on recipient-specific immune responses, and thus have inherent limitations in both sensitivity and selectivity, especially in distinguishing rejection from infection. The investigators' goal is to use a novel DNA sequencing technology to develop a rapid, inexpensive, and non-invasive method for monitoring organ transplant recipients for graft rejection. The investigators' research is driven by the fact that acute and chronic rejection of thoracic organ transplants remain major causes of patient morbidity and mortality, and require intense resource utilization. The investigators' novel approach is the first to focus on a donor-specific marker of acute rejection. The investigators will use high throughput next generation sequencing to monitor the proportion of cell-free donor DNA to recipient DNA in the recipient's blood stream as a marker of rejection. This approach is enabled by the fact that an organ transplant is also effectively a genome transplant, and by monitoring single nucleotide polymorphisms that are specific to the donor's genome (and are not shared with the recipient's genome) one can measure the relative health of the transplanted organ. The investigators' preliminary studies show that cell-free donor DNA levels in the serum of heart transplant recipients increase prior to diagnosis of acute rejection by endomyocardial biopsy, but remain at stable low levels in the absence of acute rejection.

ELIGIBILITY:
Inclusion Criteria:

1. All ages of heart or lung transplant recipients
2. Recipients of re-do heart or re-do lung transplants

Exclusion Criteria:

1. Patients wait-listed for multiple organ transplantation (e.g. heart-kidney, heart-liver, heart and lung.)
2. Unable or unwilling to return to Stanford for biopsy and follow-up procedures
3. Followed by Palo Alto VA Hospital after transplant surgery (VA patients are transplanted at Stanford, but all subsequent clinical care is performed at VA hospitals)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stanford and Lucille Packard adult and pediatric, lung or heart transplant recipients and Kaiser adult heart transplant recipients.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09-29 (Actual); Study Completion 2013-09-29 (Actual)

PRIMARY OUTCOMES:
Proportion of cell-free donor DNA to recipient DNA in the recipient's blood stream as a marker of rejection. | The outcome measure is assessed for each patient up to 5 years post-transplant. Sampling timepoints include: Days 1, 2, 3, Weeks 1, 2, 4, 6, 8, 10, 12, Months 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 and quarterly through year 5
  We will use high throughput next generation sequencing to monitor the proportion of cell-free donor DNA to recipient DNA in the recipient's blood stream as a marker of rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Khush, MD MAS FACC, Principal Investigator — Stanford University Hospital and Clinics
Locations (2):
- United States (2):
  - Kaiser Permanente Northern California, Santa Clara, California
  - Stanford University Hospital and Clinics, Stanford, California

REFERENCES:
- [Background] Snyder TM, Khush KK, Valantine HA, Quake SR. Universal noninvasive detection of solid organ transplant rejection. Proc Natl Acad Sci U S A. 2011 Apr 12;108(15):6229-34. doi: 10.1073/pnas.1013924108. Epub 2011 Mar 28. PMID 21444804
- [Result] De Vlaminck I, Khush KK, Strehl C, Kohli B, Luikart H, Neff NF, Okamoto J, Snyder TM, Cornfield DN, Nicolls MR, Weill D, Bernstein D, Valantine HA, Quake SR. Temporal response of the human virome to immunosuppression and antiviral therapy. Cell. 2013 Nov 21;155(5):1178-87. doi: 10.1016/j.cell.2013.10.034. PMID 24267896
- [Result] De Vlaminck I, Valantine HA, Snyder TM, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Bernstein D, Weisshaar D, Quake SR, Khush KK. Circulating cell-free DNA enables noninvasive diagnosis of heart transplant rejection. Sci Transl Med. 2014 Jun 18;6(241):241ra77. doi: 10.1126/scitranslmed.3007803. PMID 24944192
- [Derived] Keller M, Bush E, Diamond JM, Shah P, Matthew J, Brown AW, Sun J, Timofte I, Kong H, Tunc I, Luikart H, Iacono A, Nathan SD, Khush KK, Orens J, Jang M, Agbor-Enoh S. Use of donor-derived-cell-free DNA as a marker of early allograft injury in primary graft dysfunction (PGD) to predict the risk of chronic lung allograft dysfunction (CLAD). J Heart Lung Transplant. 2021 Jun;40(6):488-493. doi: 10.1016/j.healun.2021.02.008. Epub 2021 Feb 20. PMID 33814284
- [Derived] Agbor-Enoh S, Jackson AM, Tunc I, Berry GJ, Cochrane A, Grimm D, Davis A, Shah P, Brown AW, Wang Y, Timofte I, Shah P, Gorham S, Wylie J, Goodwin N, Jang MK, Marishta A, Bhatti K, Fideli U, Yang Y, Luikart H, Cao Z, Pirooznia M, Zhu J, Marboe C, Iacono A, Nathan SD, Orens J, Valantine HA, Khush K. Late manifestation of alloantibody-associated injury and clinical pulmonary antibody-mediated rejection: Evidence from cell-free DNA analysis. J Heart Lung Transplant. 2018 Jul;37(7):925-932. doi: 10.1016/j.healun.2018.01.1305. Epub 2018 Jan 31. PMID 29500138
- [Derived] Vollmers C, De Vlaminck I, Valantine HA, Penland L, Luikart H, Strehl C, Cohen G, Khush KK, Quake SR. Monitoring pharmacologically induced immunosuppression by immune repertoire sequencing to detect acute allograft rejection in heart transplant patients: a proof-of-concept diagnostic accuracy study. PLoS Med. 2015 Oct 14;12(10):e1001890. doi: 10.1371/journal.pmed.1001890. eCollection 2015 Oct. PMID 26466143